CLINICAL TRIAL: NCT03264456
Title: Pretreatment Staging of High-Risk Prostate Cancer With 18F-Fluciclovine PET/MRI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Samuel Joseph Galgano, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300000291
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Results first posted 2020-01-22 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18F] Fluciclovine PET/MRI (Experimental): [18F] Fluciclovine PET/MRI for pretreatment staging of high-risk prostate cancer
  Interventions: Diagnostic Test: [18F] Fluciclovine PET/MRI; Drug: [18F] fluciclovine

INTERVENTIONS:
Diagnostic Test: [18F] Fluciclovine PET/MRI — [18F] fluciclovine PET/MRI
Drug: [18F] fluciclovine — [18F] fluciclovine

SUMMARY:
There is great need for improved preoperative imaging in men with high-risk prostate cancer. Investigators propose to develop and validate an optimized simultaneous PET/MRI protocol for local, regional and whole body preoperative staging in a single imaging session using the amino acid PET tracer, F-18 fluciclovine. Despite advances in the diagnosis and treatment of prostate cancer, the preoperative staging of men with prostate carcinoma (PCa) is currently problematic. Conventional imaging is falsely negative for regional lymph node metastases in a substantial fraction of men. In particular, approximately 35% of men with high-risk prostate cancer will have biochemical recurrence even after optimal surgical resection. A major benefit of simultaneous acquisition of a multiparametric prostate MRI (mpMRI) and F-18 fluciclovine PET includes having the patient undergo a single imaging study which provides both anatomic and molecular characterization of the tumor, including metastases which would potentially be missed by conventional anatomic imaging and size criteria. Additionally, simultaneous acquisition will improve co-registration of the PET and MR data which is valuable for small lesions and in anatomically complex regions. Although the use of fluciclovine in the characterization of the primary PCa remains to be established, the anatomic detail provided by conventional mpMRI will complement the detection of small volume metastatic disease by fluciclovine PET. Additionally, the use of hybrid PET/MRI technology allows for the assessment of dynamic tracer uptake and washout during the whole body and regional PET/MRI scan, which may demonstrate the ability to increase detection of the primary PCa on fluciclovine PET. If F-18 fluciclovine PET/MRI can reliably and accurately detect nodal metastases in high-risk prostate cancer patients, surgeons may use this new technology to develop new treatment algorithms for the optimal management of these patients.

ELIGIBILITY:
Inclusion Criteria:

- High-risk biopsy-proven treatment-naïve prostate adenocarcinoma (Gleason score ≥ 8 and/or serum PSA > 20)

Exclusion Criteria:

* Inability to tolerate or undergo PET/MRI
* Previous or current hematologic or lymphatic disorder (including leukemia, lymphoma, Castleman's disease, etc.)
* Recurrent prostate adenocarcinoma
* Known visceral, osseous, or extrapelvic metastases prior to fluciclovine-PET/MRI
* Known allergy to glucagon or gadolinium-based contrast

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Galgano, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Galgano SJ, McDonald AM, Rais-Bahrami S, Porter KK, Choudhary G, Burgan C, Bhambhvani P, Nix JW, Morgan DE, Li Y, Thomas JV, McConathy J. Utility of 18F-Fluciclovine PET/MRI for Staging Newly Diagnosed High-Risk Prostate Cancer and Evaluating Response to Initial Androgen Deprivation Therapy: A Prospective Single-Arm Pilot Study. AJR Am J Roentgenol. 2021 Sep;217(3):720-729. doi: 10.2214/AJR.20.24509. Epub 2020 Oct 14. PMID 33052718

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three consented patients chose not to undergo the initial PET/MRI scan prior to the scan being performed. Additionally, one patient's images were lost to data corruption and the patient was not included in the final analysis.
Period: Overall Study
Arm/Group | [18F] Fluciclovine PET/MRI
Started | 18
Completed | 14
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | [18F] Fluciclovine PET/MRI
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 65.6 [50 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Primary Lesions Detected
Description: Number of patients with primary lesions detected on 18-F fluciclovine PET/MRI
Time Frame: Baseline through 24 hr
Measure: Count of Participants; unit: Participants
Arm/Group | [18F] Fluciclovine PET/MRI
Number analyzed (Participants) | 14
Participants | 14

2. Primary Outcome: Number of Patients With Nodal Metastases Detected on Fluciclovine-PET/MRI
Description: Number of patients with nodal metastases detected on [18F]fluciclovine PET/MRI
Time Frame: Baseline through 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | [18F] Fluciclovine PET/MRI
Number analyzed (Participants) | 14
Participants | 7

3. Secondary Outcome: Number of Patients With Nodal Metastases Detected on PET/MRI vs. MRI
Description: Compare number of patients with nodal metastases detected on [18F]fluciclovine PET/MRI to number of patients with metastases detected on prostate MRI alone.
Time Frame: Baseline through 24 hours
Population: Total number of patients who demonstrated nodal metastatic disease on fluciclovine-PET/MRI
Measure: Count of Participants; unit: Participants
Arm/Group | [18F] Fluciclovine PET/MRI
Number analyzed (Participants) | 7
Participants
  MR alone | 3
  PET/MRI | 7

4. Secondary Outcome: Follow-up
Description: Changes in primary lesion maximum SUV between pretreatment PET/MRI and followup PET/MRI following 8 weeks of androgen deprivation therapy (ADT)
Time Frame: Baseline through 8 weeks
Population: Number of patients in total cohort who underwent ADT
Measure: Mean (Standard Deviation); unit: standardized uptake values
Arm/Group | [18F] Fluciclovine PET/MRI
Number analyzed (Participants) | 10
standardized uptake values
  Pretreatment maximum SUV | 7.1 (1.7)
  Maximum SUV after 8 weeks of ADT | 3.5 (2.0)

ADVERSE EVENTS:
Time Frame: Baseline through 8 week follow-up scan
Description: Given that fluciclovine is a FDA clinically approved radiotracer with almost no risk of serious adverse events and all cause mortality, the expected risk of these in this study is effectively 0.
Arm/Group | [18F] Fluciclovine PET/MRI
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT03264456/Prot_SAP_000.pdf